CLINICAL TRIAL: NCT05115279
Title: The Surgical Outcomes of Breast Conservative Surgery for Post Chemotherapy Tumour Size in Patients Had a Favourable Response to Neoadjuvant Chemotherapy
Brief Title: Outcomes of Breast Conservative Surgery for Post Chemotherapy Tumour Size After Response to Neoadjuvant Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, samir hosny mahmoud, breast surgeon, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: assuitu faculty of medicine
Record Dates: First submitted 2021-10-07; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Safety of Excision the New Tumor Size

STUDY DESIGN:
Intervention Model Description: Type of the study: prospective descriptive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast conservative Surgury after neuadjvant chemotherapy (Other): Breast conservative Surgury
  Interventions: Procedure: breast conservative surgery for post chemotherapy tumour size

INTERVENTIONS:
Procedure: breast conservative surgery for post chemotherapy tumour size — * Skin preparation by povidine iodine.
  * Excision of the mass with safety margin.
  * Sentinel axillary lymph node or complete axillary clearance depend on axillary lymph node status
  * All specimens were oriented with sutures
  * A frozen section examination of the specimen was performed intraoperative
  * When the margin status was inadequate, a re-excision was performed
  * Closure as drawn by different oncoplastic technique

SUMMARY:
Breast cancer is the most common cancer among women. The morbidity and mortality of breast cancer are much higher than those observed with other female cancers (1). The incidence of breast cancer increases with age (2, 3). Approximately 1.7 million new cases are estimated to occur worldwide, and mortality is increasing in developing countries, primarily because the disease is not diagnosed until it is in an advanced stage(4) Neoadjuvant chemotherapy (NACT) is considered the standard of care for the management of locally advanced breast cancer and although this treatment has historically been reserved for those with inoperable breast cancer now is increasingly being used for women with earlier stage disease. (5). Encouraging results obtained with neoadjuvant chemotherapy in have resulted in clinicians using preoperative chemotherapy for patients with smaller tumors(6) . Neoadjuvant chemotherapy (NACT) could reduce surgical morbidity of the breast and axilla. By down staging of the tumor, NACT can convert patients who are candidates for mastectomy to breast-conserving surgery (BCS) candidates [7]. Furthermore, it has potential to reduce excision volumes in patients with large tumors who are already candidates for BCS. Another surgical advantage is down staging of the axilla so that axillary lymph node dissection can be avoided (8).

Complete pathological response after neoadjuvant systemic treatment is high, while complete clinical response rates are even higher. Because it is difficult to localize the original tumor bed after a complete clinical and radiological response, marking the tumor before the start of neoadjuvant systemic treatment is required to enable breast-conserving surgery afterward. Achieving adequate margins of excision is an important component of breast surgery. Local recurrence rates are significantly higher for patients who have positive margins of excision (9) some prospective and retrospective data suggested that patients with BCT after neoadjuvant therapy may have an increased risk for the development of a local recurrence .

If this were true, there would be no further advantage of neoadjuvant therapy and this treatment option could be questioned altogether.

A common question raised with respect to performing breast-conserving therapy after neoadjuvant chemotherapy is the volume of breast tissue that should be resected

DETAILED DESCRIPTION:
Study subjects:

1. Inclusion criteria:

   1. Female patients with operable breast cancer
   2. Female Patient aged from 20 to 60 years old
   3. Patients who are fit for general anesthesia.
   4. Patients who provide a written informed consent.
   5. Patient who agree to provide short term outcome data and agree to provide contact information to provide contact information.
2. Exclusion criteria:

   1. Female patients less than 20 years old
   2. Stage 4 breast cancer
   3. Patient has no pathological or clinical response to NACT
   4. Patients who are contraindicated for radiotherapy
   5. Pregnant patients in first trimester
   6. Patient with inflammatory carcinoma
3. Sample Size Calculation:

Prospective trial study include 50 patient whom fulfilled the inclusion criteria 2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): This prospective study is including patients will be diagnosed breast cancer and will receive neoadjuvant chemotherapy .

All patients underwent a preoperative clinical evaluation including physical examination (PE), ultrasonography, mammograph and MRI then biopsies of the breast tumor were performed to determine the histological subtype and receptor status Methods

Pro-operative preparation:

After confirming diagnosis of breast cancer and its molecular type patient undergoing marking the tumor and axillary lymph nodes by clips before receiving neoadjuvant chemotherapy.

Making Virtual pre-operative breast conserving surgical technique based on the previous tumor size

The Surgical steps:

* Depending on new tumor size ,site of the tumor ,breast cup size and degree of breast ptosis ;oncoplastic breast conserving technique would be selected
* A prophylactic antibiotic as first generation cephalosporin is given intravenous.
* Skin preparation by povidine iodine.
* Excision of the mass with safety margin.
* Sentinel axillary lymph node or complete axillary clearance depend on axillary lymph node status
* All specimens were oriented with sutures
* A frozen section examination of the specimen was performed intraoperative
* When the margin status was inadequate, a re-excision was performed
* Closure as drawn by different oncoplastic technique

ELIGIBILITY:
Inclusion Criteria:

* a. Inclusion criteria:

  1. Female patients with operable breast cancer
  2. Female Patient aged from 20 to 60 years old
  3. Patients who are fit for general anesthesia.
  4. Patients who provide a written informed consent.
  5. Patient who agree to provide short term outcome data and agree to provide contact information to provide contact information.

     Exclusion Criteria:Exclusion criteria:

  <!-- -->

  1. Female patients less than 20 years old
  2. Stage 4 breast cancer
  3. Patient has no pathological or clinical response to NACT
  4. Patients who are contraindicated for radiotherapy
  5. Pregnant patients in first trimester
  6. Patient with inflammatory carcinoma

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 1 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
breast conservative surgery after neoadjuvant chemotherapy | 4 years
  negative inked margin by intraoperative frozen section annual free PET CT scan from recurrence anf metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code